CLINICAL TRIAL: NCT02391246
Title: A Dual Time Point FDG-PET to Differentiate Between Recurrent Brain Tumor and Radionecrosis
Brief Title: Radionecrosis and FDG PET
Acronym: DTPI FDG-PET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Lionel Zuckier, Principal Investigator, Ottawa Hospital Research Institute
Other Study IDs: 20150094-01H
Record Dates: First submitted 2015-02-08; First posted 2015-03-18 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Malignant Glioma
Keywords: central nervous system tumours; [18F]-fluorodeoxyglucose
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Positron Emission Tomography Imaging: Dual time point imaging with 250 MBq of 18F-Fluorodeoxyglucose (18F-FDG)
  Interventions: Other: Positron Emission Tomography Imaging

INTERVENTIONS:
Other: Positron Emission Tomography Imaging — Participants will receive an intravenous injection of 250 MBq (megabecquerels) of 18F-Fluorodeoxyglucose (18F-FDG). The first Positron Emission Tomography (PET) acquisition of the head will occur one hour post-injection. The second acquisition will take place 3 hours post-injection. Both early and late PET images will be manually co-registered with the participant's most recent magnetic resonance images.

SUMMARY:
Gliomas are the most common malignant primary central nervous system (CNS) tumours. When high-grade gliomas (HGG) recur, subsequent magnetic resonance (MRI) imaging, with additional sequences is required.The Positron Emission Tomography (PET) radiotracer [18F]-fluorodeoxyglucose (FDG) will be used in this study to distinguish between changes seen on MRI which can be a reflection of pseudoprogression, radiation necrosis, or recurrence.

DETAILED DESCRIPTION:
Molecular imaging has been used to distinguish recurrent tumor from post-treatment changes through the use of positron emission tomography (PET) as well as other techniques. The best-studied PET radiotracer for this application is [18F]-fluorodeoxyglucose (FDG). Normal brain matter is very FDG-avid, making it more difficult to identify lesions and in addition, inflammation associated with radiation injury has been shown to be FDG avid.

In light of this, variations of the standard FDG protocols have been proposed in order to increase overall accuracy, including dual time point imaging (DTPI), consisting of injecting the patient with the standard radiotracer and acquiring two sets of images several hours apart, typically the normal initial images in addition to a delayed acquisition set.

There is good reason to suspect that DTPI FDG-PET would be useful a technique for characterizing lesions in the brain. It's been shown that FDG uptake by normal brain parenchyma initially increases then decreases with time, while tumor uptake typically increases and then plateaus. This pattern of increasing and then decreasing FDG activity has also been seen in inflammatory tissue. The difference in FDG uptake at different times is what allows for a better distinction between malignant and benign tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Able and willing to comply with the study procedures
* The patient must be followed at The Ottawa Hospital for a tissue-proven, grade III or IV glioma.
* The patient must have been treated in the past with radiotherapy for glioma.
* A disease recurrence is suspected based on clinical symptoms and/or imaging results.

Exclusion Criteria:

* Missing information regarding tumor type and grade
* Brain biopsy in the ten days preceding DTPI FDG-PET
* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients who have previously been treated with radiochemotherapy for high grade gliomas who are clinically assessed with a brain MRI for suspected disease recurrence.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity percentages | 3 years
  The sensitivity and specificity of dual time point imaging (DTPI) FDG-PET/CT will be compared to the sensitivity and specificity of MR imaging obtained as standard of care for identifying glioma recurrence post-treatment.

SECONDARY OUTCOMES:
Cost efficiency analysis | 3 years
  At the conclusion of the trial, a cost-efficiency analysis will be performed in an attempt to determine an optimally accurate and cost-efficient imaging strategy for the diagnosis of glioma recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel S Zuckier, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada